CLINICAL TRIAL: NCT06630312
Title: Glycemic Response of Whole Beans and Bean Products
Acronym: BH-GLY
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Donna Winham, Associate Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 22-375-00; 58-5050-8-009 (Other Grant/Funding Number: USDA/ARS - Pulse Crop Health Initiative)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Body Mass Index, Normal; Postprandial Hyperglycemia
Keywords: Normoglycemia; Glucose, postprandial; Insulin; alpha galactosidase; young adults
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance | interventions — alpha-Galactosidase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Yellow beans (Placebo Comparator): Yellow beans, cooked in spaghetti sauce
  Interventions: Dietary Supplement: Placebo
- Yellow beans with AGS (Experimental): Yellow beans, cooked in spaghetti sauce, with AGS treatment
  Interventions: Dietary Supplement: Alpha galactosidase
- Yellow bean pasta (Placebo Comparator): Yellow bean pasta with spaghetti sauce
  Interventions: Dietary Supplement: Placebo
- Yellow bean pasta with AGS (Experimental)
  Interventions: Dietary Supplement: Alpha galactosidase

INTERVENTIONS:
Dietary Supplement: Alpha galactosidase — Alpha galactosidase capsule, 600 GALU, manufacturer Equate brand, Walmart. Powder contents from one capsule were stirred into 16 g spaghetti sauce and served before the main meal.
  Other Names: Beano
  Arms: Yellow bean pasta with AGS; Yellow beans with AGS
Dietary Supplement: Placebo — Placebo is 16 gm of spaghetti sauce served before the meal in a condiment cup. It is the same set up as the intervention except the 'intervention' contains the AGS.
  Arms: Yellow bean pasta; Yellow beans

SUMMARY:
The main goal of this clinical trial is to learn if alpha-galactosidase (tradename Beano) changes in post-prandial (after-meal) blood glucose after eating whole cooked whole pulses or pulse-based pasta products in comparison to the same foods without alpha-galactosidase. Comparison of postprandial blood insulin and triglyceride levels, appetite, and gastrointestinal symptoms of flatulence, bloating, and stool changes will be evaluated by comparisons of the alpha-galactosidase and the pulse form (whole vs. pasta). In addition to blood glucose, such as flatulence and bloating, postprandial glucose, insulin, and appetite of individuals.

The study design is a 4x4 crossover and the population is healthy volunteers aged 21-34 with normal glucose response and body weight.

The primary hypothesis is that alpha-galactosidase will cause increased postprandial blood glucose for both whole and pasta pulse foods. The secondary hypothesis is that gastrointestinal symptoms will be less for both meals with the alpha-galactosidase. Other comparisons are exploratory.

Participants will come in fasting for one morning per week and receive the food treatments in randomized order. Test measurements will be taken over a four hour period.

DETAILED DESCRIPTION:
The 4 test treatments (yellow whole bean, yellow whole bean and alpha-galactosidase (AGS), yellow bean flour pasta, yellow bean flour pasta and AGS) will be administered in semi-randomized order once every four weeks. Participants will be randomized to whole beans or bean pasta, and within the meal group randomized again to receive the AGS treatment or not. Pulses will be served with a standardized amount of spaghetti sauce. The treatment intervention consisted of 16 gm of pasta sauce with either no AGS or 600 GALU of AGS.

The test participants were required to consume the entire test meal in 7-9 minutes while being observed. Venous blood samples were collected for blood glucose and insulin levels at time 0 (fasting) and at 30, 60, 90, 120, and 180 minutes post treatment (timing of the post-treatment draws started at time 0 [post-treatment], which is when the participant finishes consuming the treatment meal). Triglycerides were measured at time 0, 60, 120, 180 minutes post-treatment.

Blood samples were processed according to laboratory instructions and sent out for analysis by Quest Diagnostics. Breath hydrogen samples were collected at times 0 (fasting), 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, and 180 minutes post treatment. Samples were measured at the end of the 4-hour test period in sequential order on the same calibrated instrument.

Anthropometric measures of weight, height, waist circumference, and blood pressure were collected at screening and weight, waist circumference, and blood pressure will be collected at the start of each test day. Thirteen hours before testing, participants will consume a standardized frozen meal to reduce the potential variation in glycemic responses on test day due to varying pre-evening dietary intakes. This control meal was selected by each participant before the start of the study. Each participant was provided the same frozen meal every time, since the subjects serve as their own controls. The day before test day, participants completed a 24-hour food recall, satiety, and gastrointestinal questionnaires .

During each test day participants completed satiety questionnaires, sensory questionnaires, and a gastrointestinal questionnaire. Satiety questionnaires were completed every 45 minutes after the first bite. The sensory questionnaire was completed immediately following the entire test meal being eaten. The gastrointestinal questionnaire was completed the evening before the test day, at 165 minutes following the first bite of the test meal, the evening of testing, and the following evening.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20-29.9 kg/m2
* Height range of 60-74"
* HbA1C between 4.9-5.7%
* Individuals who consumed breakfast on most days
* Women who were not pregnant or lactating
* Individuals who could walk and eat independently
* Individuals who were willing to eat beans and bean pasta
* Individuals who were willing to restrict moderate and vigorous exercise, caffeine, alcohol, or herbal teas for 24 hours prior to testing

Exclusion Criteria:

* Persons who smoke cigarettes, tobacco of other kinds or e-cigarettes
* Vegetarian/Vegan
* Uncontrolled health conditions and/or diagnosis of gastrointestinal disease
* Intake of any medications and/or dietary supplements affecting glucose levels
* Individuals with HbA1C level >5.9% at screening
* Individuals with an allergy to legumes, tomatoes, nus, wheat, or gluten
* Known latex allergy
* Known allergy to mold or alpha-galactosidase enzyme products
* Never had blood drawn before from arm
* Known difficulty with blood draws, e.g., feeling faint, or dizzy
* Individual who have had a recent weight gain or loss (>10% over 6 months)
* Persons who work altered shifts
* Abnormal score on the Three-Factor Eating Questionnaire
* Unwillingness or inability to follow study protocol

Ages: 21 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men, Women
Enrollment: 21 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose | Time 0 (fasting), then every 30 minutes for 3 hours
  Venous blood sample of glucose

SECONDARY OUTCOMES:
Postprandial insulin | Time 0 (fasting), then every 30 minutes for 3 hours
  Venous blood sample of insulin
Postprandial triglycerides | Time 0 (fasting), then every 60 minutes for 3 hours
  Venous blood sample of triglycerides
Satiety or Appetite evaluation | Time 0 (fasting), then 45 minutes post-ingestion, and 30 minutes after that for seven data points
  Participant completion of satiety and appetite ranking survey. Satiety level measured using a visual analog scale (0-100). A higher score indicates greater satiety.
Breath hydrogen | Time 0 (fasting), then every 15 minutes for 3 hours
  Participants blew into Quintron & Easy Sampler device for breath hydrogen measures before testing, and post-ingestion of the test meal for 3 hours.
Gastrointestinal symptoms | Pre-test day, evening of testing in the am, and evening on the day after testing
  Participants completed symptom check list for flatulence, bloating, belching, and the Bristol Stool chart for the pre-test day, evening after testing, and post-test day.

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
I am willing to share if I am asked about it. I do not plan to upload to a data repository at this time.